CLINICAL TRIAL: NCT02467816
Title: Technology and Design Innovation to Support 21st Century School Nutrition
Brief Title: Technology and Design Innovation for School Lunch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: University of California (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014-12-7010
Record Dates: First submitted 2015-06-08; First posted 2015-06-10 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Childhood Obesity
Keywords: Secondary schools; School lunch; Plate waste
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- School lunch intervention (Experimental): Intervention schools (6 middle and 6 high) will receive the complete school lunch intervention for two school years.
  Interventions: Behavioral: SmartMeal application; Behavioral: Distributed points of sale; Behavioral: Staff wellness curriculum
- School lunch control (No Intervention): Control schools (6 middle and 6 high) will not receive the school lunch intervention for two school years. Lunch delivery will proceed as normal.

INTERVENTIONS:
Behavioral: SmartMeal application — The SmartMeal application is a smartphone application that will allow students to pre-order school meals, receive nutrition information about school meals, and provide feedback about school meals to Student Nutrition Services.
  Arms: School lunch intervention
Behavioral: Distributed points of sale — To increase points of sale for school meals (outside the cafeteria), school meals will be sold at hot and cold mobile food carts and vending machines throughout the school.
  Arms: School lunch intervention
Behavioral: Staff wellness curriculum — A wellness curriculum will be implemented that encourages teachers and staff members to eat school meals and promote them to students.
  Arms: School lunch intervention

SUMMARY:
This study will evaluate an innovative school lunch intervention that is designed to increase school meal participation and improve dietary intake among middle and high school students.

DETAILED DESCRIPTION:
Improving dietary intake among low-income youth is critical to reducing obesity, and schools are arguably the most important system in which to intervene. In 2010, Congress passed the Healthy, Hunger-Free Kids Act to better align school meal standards with the Dietary Guidelines, making school meals a nutritious option for students. Increasing participation in the school meal program, therefore, especially among low-income youth, has the potential to improve dietary intake among students and ultimately reduce childhood obesity.

Over three school years, the University of California (Berkeley's School of Public Health and the Division of Agriculture and Natural Resources' Nutrition Policy Institute) will evaluate an innovative, student-centered school-lunch intervention to increase school lunch participation and improve dietary intake among low-income middle and high school students. The project will be conducted in the San Francisco Unified School District (SFUSD), a large and diverse urban district serving over 32,000 students (70% of total) eligible for free or reduced-price meals. The intervention, developed in partnership with the global design firm IDEO, aims to promote healthier habits by leveraging principals of behavior economics. The intervention involves the following three components: 1) a smartphone application (SmartMeal) that allows students to pre-order school lunches, receive nutrition information about school lunch options, and provide feedback about meals to food service staff, 2) distributed points of sale for school meals, achieved through the addition of mobile food carts and vending machines, and 3) a staff wellness curriculum that encourages staff to promote school meals and model healthful eating behaviors to students.

ELIGIBILITY:
Inclusion Criteria:

* All 7th-10th grade students at participating schools are eligible to participate in the student survey
* All 6th-12th grade students who eat the school lunch are eligible to participate in plate waste data collection
* All 7th-10th grade teachers are eligible to participate in the teacher survey

Exclusion Criteria:

* There are no exclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 27406 (Actual)
Dates: Start 2016-02; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change in school lunch participation | 2 years
  Daily school lunch participation records broken down by grade, gender, and free or reduced-price meal eligibility at each school.

SECONDARY OUTCOMES:
Change in plate waste during lunch among students who eat school lunch | 2 school years
  Individual-level waste of food components achieved through visual estimation and aggregate waste of food components achieved through weighing.
Change in fruit consumption at lunch | 2 school years
  Student survey that asks about fruits consumed at lunch yesterday
Change in vegetable consumption at lunch | 2 school years
  Student survey that asks about vegetables consumed at lunch yesterday
Change in weekly fruit consumption | 2 school years
  Student survey that asks about fruits consumed during a typical week
Change in weekly vegetable consumption | 2 school years
  Student survey that asks about vegetables consumed during a typical week
Change in variety of fruits consumed by students at lunch | 2 school years
  Student survey that asks about fruits consumed at lunch yesterday
Change in variety of vegetables consumed by students at lunch | 2 school years
  Student survey that asks about vegetables consumed at lunch yesterday
Change in variety of fruits consumed by students each week | 2 school years
  Student survey that asks about fruits consumed during a typical week
Change in variety of vegetables consumed by students each week | 2 school years
  Student survey that asks about vegetables consumed during a typical week
Change in body mass index (index) | 2 school years
  BMI data collected each year on 7th and 9th grade students via the California Physical Fitness Test

CONTACTS AND LOCATIONS:
Overall Officials: Kristine A Madsen, MD MPH, Principal Investigator — University of California, Berkeley; Lorrene Ritchie, PhD RD, Principal Investigator — University of California Division of Agriculture and Natural Resources
Locations (24):
- United States (24):
  - Academy High School and Ruth Asawa School of the Arts, San Francisco, California
  - AP Giannini Middle School, San Francisco, California
  - Aptos Middle School, San Francisco, California
  - Balboa High School, San Francisco, California
  - Burton High School, San Francisco, California
  - Everett Middle School, San Francisco, California
  - Francisco Middle School, San Francisco, California
  - Galileo High School, San Francisco, California
  - Herbert Hoover Middle School, San Francisco, California
  - James Denman Middle School, San Francisco, California
  - James Lick Middle School, San Francisco, California
  - John O'Connell High School, San Francisco, California
  - June Jordan High School, San Francisco, California
  - Lincoln High School, San Francisco, California
  - Lowell High School, San Francisco, California
  - Marina Middle School, San Francisco, California
  - Marshall High School, San Francisco, California
  - Martin Luther King Middle School, San Francisco, California
  - Mission High School, San Francisco, California
  - Presidio Middle School, San Francisco, California
  - Roosevelt Middle School, San Francisco, California
  - Visitacion Valley Middle School, San Francisco, California
  - Wallenberg High School, San Francisco, California
  - Washington High School, San Francisco, California